CLINICAL TRIAL: NCT02491918
Title: Visual Axis Obscuration and Postoperative Complications Following Pediatric Cataract Surgery With Introacular Lens Implantation In-the-bag Versus Posterior Optic Capture : A Randomized, Clinical Trial
Brief Title: Clinical Trial : Complications of in the Bag IOL Versus Optic Capture of IOL in Pediatric Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, Director, Iladevi Cataract and IOL Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-009; 2013 Research Foundation Grant (Other Grant/Funding Number: ASCRS Foundation Research Grant)
Record Dates: First submitted 2015-06-29; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Posterior Capsule Opacification; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Cataract Extraction; Lens Implantation, Intraocular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In the bag IOL (Active Comparator): Cataract surgery with IOL implantation in the capsular bag
  Interventions: Procedure: cataract surgery; Procedure: Intraocular lens implantation
- Optic Capture of IOL (Active Comparator): intraocular lens implantation in the capsular bag with posterior optic capture
  Interventions: Procedure: cataract surgery; Procedure: Intraocular lens implantation

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery in children
Procedure: Intraocular lens implantation — intraocular lens implantation in the capsular bag or optic capture

SUMMARY:
This prospective, randomized, clinical trial looks to compare children undergoing congenital cataract surgery with intraocular lens (IOL) implantation in terms of visual axis obscuration as well as postoperative complications such as glaucoma, inflammation and IOL centration when IOL fixation is performed using two different techniques : 1) conventional in the bag IOL implantation with anterior vitrectomy, and, 2) posterior optic capture of the IOL through the posterior capsulorhexis without any vitrectomy. 61 eyes of 61 children randomized to receiving IOL implantation using one of the two techniques will be followed up until 12 months postoperatively.

DETAILED DESCRIPTION:
This prospective, randomized, controlled, clinical trial compares visual axis obscuration as well as intra and postoperative complications in children undergoing cataract surgery with IOL implantation using one of two techniques :

1. in the bag IOL with limbal anterior vitrectomy
2. posterior optic capture of IOL optic through the posterior capsulorhexis without any vitrectomy.

The aim is to evaluate whether avoiding anterior vitrectomy is a feasible option, particularly younger children, where anterior vitrectomy has become an integral part of the routine surgical strategy.

All children will be evaluated at 1 month, 3 months, 6 months and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated cataract,
* unilateral or bilateral cataract,
* corneal diameter >9.0mmHg

Exclusion Criteria:

* pre-existing glaucoma,
* uveitis,
* ocular comorbidity,
* microphthalmos,
* microcornea,
* parents not consenting to participate in study,
* traumatic cataract

Ages: 15 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Posterior capsule opacification requiring surgery | 12 months postoperatively
  opacification of visual axis

SECONDARY OUTCOMES:
inflammation on slitlamp examination | 12 months postoperatively
  cell depostis
inflammation on slitlamp examination | 12 months postoperatively
  posterior synechiae
intraocular pressure in mmHg | 12 months postoperatively
  glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: abhay vasavada, MS,FRCS, Study Director — Iladevi Cataract & IOL Research Centre, Ahmedabad, India